CLINICAL TRIAL: NCT05988281
Title: The Success of Implant Supported Restorations After Immediate Implant Placement or Delayed Implant Placement With or Without Ridge Preservation
Brief Title: Success of Implant Restorations After Immediate or Delayed Implant Placement With/Without Ridge Preservation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital General Universitario Morales Meseguer (Other)
Responsible Party: Principal Investigator, Ruben Garcia-Sanchez, Dr. Ruben Garcia-Sanchez. Senior Lecturer., Hospital General Universitario Morales Meseguer
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UM-RP001
Record Dates: First submitted 2023-07-21; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Dental Implant

STUDY DESIGN:
Intervention Model Description: This is a prospective, parallel-group, randomized study. This study will include three groups:
  i. Immediate dental implant placement with autogenous connective tissue graft (type I).
  ii. Early dental implant placement (type II). iii. Delayed/late dental implant placement in socket-preserved sites (type III/IV).
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigator and outcome assessor will be blinded regarding group allocation as patients' ID and group will be anonimysed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Type I dental implant placement. (Experimental): Type I dental implant placement (immediately after extraction)
  Interventions: Procedure: Type I Dental implant placement.
- Type II dental implant placement. (Experimental): Type II dental implant placement (6-8 weeks after extraction)
  Interventions: Procedure: Type II Dental implant placement.
- Type III/IV placement. (Experimental): Type III/IV placement in socket preserved sites after 3-6 months.
  Interventions: Procedure: Type III/IV dental implant placement.

INTERVENTIONS:
Procedure: Type I Dental implant placement. — Placement of dental implant.
  Arms: Type I dental implant placement.
Procedure: Type II Dental implant placement. — Placement of dental implant.
  Arms: Type II dental implant placement.
Procedure: Type III/IV dental implant placement. — Placement of dental implant.
  Arms: Type III/IV placement.

SUMMARY:
The study aims to compare clinical, radiographic, patient-reported outcomes (PROMs) and cost analysis outcomes in type I, II and socket preserved sites (III/IV) implant placement at 1-year post-loading in all groups.

DETAILED DESCRIPTION:
This is a prospective, parallel-group, randomized study aiming to compare clinical, radiographic, PROMS and health-economic outcomes of type I, type II and type III/IV (in socket preserved areas) implant placement.

This study included three groups:

i. Immediate implant placement + aputogenous connective tissue graft (CTG) (type I).

ii. Early implant placement (type II, after 6-8 weeks). iii. Delayed/late placement in socket-preserved sites (type III/IV, after 3-6 months).

Up 75-90 adult, systemically healthy patients will be recruited mainly in the new patient and follow-up implant clinics which run every week at the Murcia University Dental Hospital Morales Meseguer. In addition, patients with unrestorable maxillary premolars, canines and incisors will be recruited from other relevant clinics within the same hospital, such as Periodontics, Endodontics/Dental Trauma Restorative Dentistry, Oral Surgery and Hypodontia outpatient clinics. Flyers advertising the study will also be placed in the Hospital and in the reception area to be visible.

After screening patients, the potentially eligible participants will be given the patient information sheet and they will be invited to attend the enrolment visit at Murcia University Dental Hospital Morales Meseguer . Before any study-related intervention is performed, informed consent will be obtained. During the enrolment visit, a detailed medical history will be taken and the periodontal parameters adjacent to the tooth to replace will be recorded. The GDP will be sent a letter to inform him/her about the enrolment of their patient in the study and about the need for any dental treatment (if needed).

Below is a summary of all study visits for each study group:

1. For type-I placement:

   Visit 1: Screening and oral hygiene improvement, non-invasive imaging baseline (intraoral scanning, pre-extraction CBCT) and impressions for temporary replacement.

   Visit 2: Extraction, CBCT post extraction and provision of immediate implant. Visit 3: Suture removal. Visit 4: Provision of second stage surgery after 12-14 weeks. Visit 5: Impressions for temporary restoration after 2 weeks. Visit 6: Provision of temporary restoration after 2-4 weeks. Visit 7: Impressions for final restoration after 3-6 months. Visit 8: Provision of final implant restoration. Visit 9: Final visit for data collection at 12 months post-loading and CBCT.
2. For type-II placement:

   Visit 1: Screening and oral hygiene improvement, non-invasive imaging baseline (intraoral scanning, pre-extraction CBCT) and impressions for temporary replacement.

   Visit 2: Extraction, CBCT post extraction. Visit 3: Suture removal after 1-2 weeks. Visit 4: Provision of type II placement after 6-8 weeks. Visit 5: Suture removal after 1-2 weeks. Visit 6: Provision of second stage surgery after 12-14 weeks. Visit 7: Impressions for temporary restoration after 2 weeks. Visit 8: Provision of temporary restoration after 2-4 weeks. Visit 9: Impressions for final restoration after 3-6 months. Visit 10: Provision of permanent implant restoration. Visit 11: Final visit for data collection at 12 months post-loading and CBCT.
3. For socket-preserved sites with type-III/IV placement:

Visit 1: Screening and oral hygiene improvement, non-invasive imaging baseline (intraoral scanning, pre-extraction CBCT) and impressions for temporary replacement.

Visit 2: Extraction, CBCT post extraction and provision of ARP. Visit 3: Suture removal after 1-2 weeks. Visit 4: Visit 5: Provision of type III/IV placement after 12-24weeks. Visit 5: Suture removal after 1-2 weeks. Visit 6: Provision of second stage surgery after 12-14 weeks. Visit 7: Impressions for temporary restoration after 2 weeks. Visit 8: Provision of temporary restoration after 2-4 weeks. Visit 9: Impressions for final restoration after 3-6 months. Visit 10: Provision of final implant restoration. Visit 11: Final visit for data collection at 12 months post-loading and CBCT.

ELIGIBILITY:
Inclusion Criteria:

i) Patient must have willingness to read and sign a copy of the Informed Consent Form Males and females, ≥23 years old.

ii) Patient in need of a single permanent tooth extraction with clinical and/or radiographic evidence of unrestorable maxillary premolars, canines, or incisors with at least one adjacent tooth present, and with periodontal attachment preserved at least for two thirds of the root not associated with acute periapical pathology.

iii) Post-extraction alveolar bone defect with ≤50 % buccal bone loss. This will be confirmed at Visit 2 after extraction. In case of >50% buccal bone loss, the participant will be withdrawn from the study.

iv) Patient in good general health as documented by self-assessment. v) Full mouth bleeding and plaque scores (FMBS <10% and FMPS <30%) recorded within the previous 8 weeks.

Exclusion Criteria:

i) Uncontrolled or untreated periodontal disease. ii) History of local (head and neck) radiation therapy. iii) Presence of oral lesions in the area of the extraction (such as ulceration, malignancy).

iv) Severe bruxing or clenching habits. v) Acute endodontic lesion in the test tooth or in the neighbouring areas to the extraction procedure (sites with presence of an asymptomatic chronic lesion are eligible).

vi) Medical history that includes uncontrolled diabetes or hepatic or renal disease, or other serious medical conditions that can impact on bone metabolism (e.g. rheumatoid arthritis, osteoporosis) or transmittable diseases (e.g. AIDS).

vii) History of alcohol or drug abuse. viii) Smokers. ix) Self-reported pregnancy or lactation (this criterion is due to oral tissue changes related to pregnancy and nursing which can affect interpretation of study results).

x) Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with trial participation or investigational product administration or may interfere with the interpretation of trial results and, in the judgement of the investigator, would make the subject inappropriate for entry into this trial.

xi) Malocclusion, or collapse of the occlusal vertical dimension leading to dentoalveolar compensation which could interfere with ridge preservation dimensions and measurements.

xii) Lack of adjacent sound restored or unrestored teeth.

Min Age: 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Combined success rate criteria. | 12 months after delivery of implant restoration.
  This is the success criteria described by Ong et al. 2008, in combintation with predetermined scores for PES/WES as decribed in Garcia-Sanchez et al. 2021.

SECONDARY OUTCOMES:
Pre-treatment outcome. Total Need for further bone augmentation. | At implant placement.
  Expressed as a percentage (%) of implants that required further ridge augmentation procedures during implant placement.
Pre-treatment outcome. Alveolar ridge dimensions clinically. | Immediately after dental extraction for type I, at month 2 for type II, at month 4 for type III/IV and at second stage surgery (10-12 weeks after implant placement) for all groups.
  i. Width at mesial/mid/ distal site ii. Height (from the CEJ of neighbouring teeth) at mesial /mid / distal site (clinical) at post extraction, 2 months for typeII, 4 months for Type III/IV, at second stage for all groups.
  iii. Defect characterisation.
Pre-treatment outcome. Alveolar ridge dimensions radiographic: | Immediately after dental extraction for type I, at month 2 for type II, at month 4 for type III/IV and at 12 months post-loading for all groups.
  i. Width at mesial/mid/ distal site ii. Height (from a radiopaque stent) at mesial /mid / distal site. iii. Area at post extraction, at month 2 for type2, at month 4 for Type III/IV , at 12 months post loading for all groups.
Pre-treatment outcome. Periodontal phenotype | Before dental extraction.
  This to be descibed as per EFP/AAP workshop.
Pre-treatment outcome. Keratinised attached gingivae before extraction. | Before dental extraction.
  Expressed in mm and measured with periodontal probe/photograph.
Pre-treatment outcome. Thickness of buccal wall (radiographic) before extraction. | Before dental extraction
  As measured in CBCT
Pre-treatment outcome. Soft tissue thickness buccally. | Before dental extraction.
  Either clinical or radiographic at 3mm from CEJ. Expressed in mm and measured with periodontal probe.
Pre-treatment outcome. Soft tissue recession. | Before dental extraction
  Cemento Enamel Junction/Stent as a reference point expressed in mm and measured with periodontal probe/photograph.
Pre-treatment outcome. Sounding of soft tissue vertical at proximal sites. | Before dental extraction and at implant placement.
  Expressed in mm and measured with periodontal probe.
Implant-related outcome. Survival at 12 months post-loading. | At 12-months post-loading.
  Implants still in mouth regardless of condition
Implant-related outcome. Feasibility of implant placement. | At implant placement.
  Expressed as percentages (%) of implants placed with satisfactory primary stability (> 30N/cm).
Implant-related outcome. Final torque placement. | At implant placement.
  Expressed as n/cm
Implant-related outcome. Need for further soft tissue augmentation (soft tissue contour deficiencies). | At implant placement or second stage surgery (10-12 weeks after dental implant placement).
  Expressed as percentages (%) of implants placed that requires additional soft tissue grafting.
Implant-related outcomes. Total surgical hours. | Overall surgical time in that specific arm group.
  Number of hours/minutes needed to complete specific surgical procedure.
Implant-related outcome. Papillary Fill Index | At 1 and 12 months post-loading.
  As per index agreed.
Implant-related outcome. Proximal bone levels (radiographic) | At 1 and 12 months post-loading.
  Expressed as mm of bone loss (-) /gain (+).
Implant-related outcome. Probing pocket depth around implants. | At 1 and 12 months post-loading.
  Expressed in mm after gentle probing (30-40 newtons).
Implant-related outcome. Intra - surgical complications. | At dental implant placement
  Expressed as percentage (%) of implants experiencing complications during implant placement.
Implant-related outcome. Post-surgical complications. | Period from implant placement to implant loading. Normally this period last between 10-12 weeks.
  Percentage (%) of implants experiencing complications from the moment implant was placed until loading.
Implant-related outcome. Technical/ mechanical complications | At 1 and 12 months post-loading.
  Percentage (%) of implants experiencing aforementioned complications during at 1 at 12M post Loading.
Implant-related outcome. Biologic complications. | At 1 and 12 months post-loading.
  Percentage (%) of implants experiencing aforementioned complications during at 1 at 12M post Loading.
Implant-related outcome. Post-operative clinical measurements. | Immediately after extraction and at 12 month post-loading
  i. Keratinised attached Mucosa around the implant at 12 months post loading ii.Soft tissue thickness buccally (12 months post loading -either clinical or radiographic at 3/ 5mm from implant shoulder ).
  iii. Recession. iv. Soft tissue vertical at proximal sites at 12 months post-loading. v. Changes in the external alveolar ridge contour/soft tissue (optical scan measurements). before extraction, before implant placement, and at 12 months post-loading vi. Buccal & palatal plate dimensions (height and thickness) immediately after dental extraction.
Implant-related outcome.Histomorphometry of new bone formation in type III/IV implant placement. | At 3 months of healing at the dental implant group III/IV.
  This assessed with Scanning Electron Microscope (SEM) and X-ray microtomography (XMT), to calculate the percentages of new bone within bone core samples.
Patient-reported outcome. VAS pain score after surgery for each group. | 2 weeks after implant placement surgery.
  Visual Analog Scale (VAS) divided in ten equal segments in which patient will rate pain from no pain (0) to the most severe pain that could be experienced (10).
Patient-reported outcome. Patient satisfaction with treatment outcome. | At 12 months post-loading.
  Questionnarie

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Pardo Zamora, Dr., Study Director — Universidad de Murcia. Associate Professor.; Ruben Garcia-Sanchez, Dr., Principal Investigator — Universidad de Murcia. Associate Professor.

IPD SHARING:
Plan to Share IPD: Yes
Datasets generated during and/or analysed during the current study are/will be available upon request from Dr. Guillermo Pardo Zamora (gparza@um.es). This data will become available once the study results are published. The data available will be all of the individual participant data collected during the trial, after deidentification. This data will be available 3 months after publication and ending 5 years following article publication. This data will be shared with investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose. The data will be shared to achieve the aims in the approved proposal. Proposals should be directed to Dr Guillermo Pardo Zamora (gparza@um.es). To gain access, data requestors will need to sign a data access agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 3 months after publication and ending 5 years following article publication.
Access Criteria: This data will be shared with investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose. The data will be shared to achieve the aims in the approved proposal.